CLINICAL TRIAL: NCT00082420
Title: Retinol Equivalence of Plant Carotenoids in Children
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Other Study IDs: RETEQ (completed); DK60021; NCT00072696 (obsolete NCT alias)
Record Dates: First submitted 2004-05-06; First posted 2004-05-12 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Vitamin A Deficiency
Keywords: Vitamin A malnutrition; low vitamin A status
MeSH Terms: conditions — Vitamin A Deficiency

STUDY DESIGN:
Observational Model: Case-Only

SUMMARY:
To determine vitamin A value of beta-carotene in oil capsule, spinach, and golden rice.

The experiments will be conducted in children (ages 7-9) with/without adequate vitamin A nutrition. As plant provitamin A carotenoids are a major and safe vitamin A source for a vast population in the world, it is essential to determine the efficiency of provitamin A carotenoid (mainly ß-C) conversion to vitamin A. By introducing ß-C into rice endosperm, Golden Rice may directly benefit consumers by providing vitamin A nutrition. Our investigation uses hydroponically grown, deca-deuterium labeled spinach and Golden Rice, synthetic ß-C-d10 and a vitamin A isotope reference, deca-deuterated retinyl acetate (RAc-d10), to evaluate the bioavailability and the bioconversion of plant provitamin A carotenes to retinol as compared with ß-C in oil capsules in vivo.

Our objectives will be to test the following hypotheses and to make the following determinations: (1) The absorption and bio-conversion of provitamin A carotenes taken by children are different between spinach, Golden Rice, and ß-C in oil capsules. (2) The absorption of provitamin A carotenes and their bioconversion to vitamin A are different in children with or without adequate vitamin A nutrition. (3) To define the vitamin A equivalence(s) of dietary spinach, Golden Rice, and a ß-C in oil dose by using an isotope reference method in children with or without adequate vitamin A nutrition and to compare those values with values derived from model based compartmental analysis. (4) To determine the number and time of blood samples needed for future studies in various field settings on the retinol equivalence of a large number of plant sources.

This study will be of importance in planning vitamin A deficiency prevention strategies and also will provide useful information regarding the potential efficacy of a bioengineered crop to provide vitamin A nutrition.

DETAILED DESCRIPTION:
Seventy-two children each will take two meals, lunch and supper, containing equal amounts of ß-C in labeled spinach (along with white rice), or Golden Rice (along with light colored vegetables), or ß-C oil capsules (along with white rice and light colored vegetables), every day for 7 days. Before the two meals, the volunteers will take a breakfast with a RAc-d10 dose as a reference for 7 days. The enrichment of labeled ß-C and labeled retinol in human circulation will be determined using advanced liquid chromatography / mass spectrometry and gas chromatography / mass spectrometry. Through the applications of these novel technologies, we will be able to determine the relative biological activities of endogenous carotenoids; that is, the vitamin A value of spinach, Golden Rice, and ß-C in oil capsules for children with/without vitamin A malnutrition.

ELIGIBILITY:
Inclusion Criteria:

* 7-9 years old

Exclusion Criteria:

* Parasitic infection

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: healthy children with normal or marginal vitamin A nutrition
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2004-09; Study Completion 2005-11 (Actual)

REFERENCES:
- [Background] Li L, Wang Y, Wu J, Zhu R. [Bioefficacy of plant carotenoid to vitamin A in school age children]. Wei Sheng Yan Jiu. 2007 Sep;36(5):547-51. Chinese. PMID 18095563
- [Result] Lei Li, Yin Wang, Shi-an Yin, Michael A Grusak, Robert M Russell, Guangwen Tang. Bioconversion of spinach β-carotene in Chinese children with noemal or marginal vitamin A status. FASEB J. 2006 20:A1319